CLINICAL TRIAL: NCT05498324
Title: External Validation of the 4C Mortality Score for Hospitalised Patients With COVID-19 in a Tunisian Cohort
Acronym: 4C
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Other Study IDs: 4C Score
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: COVID-19 Pandemic
Keywords: covid-19; SARS-COV2; 4c score; validation
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Risk prediction scores are important tools to support clinical decision-making for patients with coronavirus disease (COVID-19). The objective of this paper was to validate the 4C mortality score, originally developed in the United Kingdom, for a tunisian population, and to examine its performance over time.

DETAILED DESCRIPTION:
Coronavirus disease (COVID-19) caused by the Severe Acute Respiratory Syndrome Virus 2 (SARS-CoV-2) can progress to acute respiratory distress syndrome, multiorgan failure, and death in some cases. The clinical presentation and progression of COVID-19 in patients is highly variable, which makes it difficult for clinicians to triage patients and determine their prognostic risk. A simple, validated prognostic tool using data that is available at presentation can help clinicians better prognosticate and support clinical decision-making . Numerous tools to predict mortality in COVID-19 patients have been developed, but many are limited due to small derivation cohort sizes and/or inadequate validation.

The 4C mortality score is an accessible risk stratification score developed by the International Severe Acute Respiratory and Emerging Infections Consortium (ISARIC). It was derived and internally validated on a large, diverse cohort within the United Kingdom but requires external validity to confirm its generalizability.

The objective of this study was to validate the 4 C Mortality risk score to predict in-hospital mortality among adults hospitalised with COVID-19 in a Tunisian cohort.

.

ELIGIBILITY:
Inclusion Criteria:

* patients ≥18 years old
* admitted to one of the participating hospitals with a confirmed case of COVID-19 defined by a positive reverse transcriptase-PCR (RT-PCR) assay of a nasopharyngeal swab associated with compatible clinical manifestations

Exclusion Criteria:

* under the age of 18
* Incomplete electronic records were excluded from the analysis.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in this study had a positive SARS-CoV-2 PCR test result and were admitted through the emergency department one of the participating centers, between november 1st,2020 to December 1st, 2021.
Sampling Method: Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
The primary outcome was all-cause in-hospital mortality rate | 30 days after inclusion
  The primary outcome was all-cause in-hospital mortality rate

SECONDARY OUTCOMES:
ICU admission rate | 30 days after inclusion
  ICU admission rate
combined outcome | 30 days after inclusion
  all-cause in-hospital mortality and/or ICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Bel Haj Ali Khaoula, MD, Study Director — CHU Fattouma Bourguiba Monastir, service des urgences
Locations (1):
- Fattouma Bourguiba University Hospital, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gordon AJ, Govindarajan P, Bennett CL, Matheson L, Kohn MA, Camargo C, Kline J. External validation of the 4C Mortality Score for hospitalised patients with COVID-19 in the RECOVER network. BMJ Open. 2022 Apr 21;12(4):e054700. doi: 10.1136/bmjopen-2021-054700. PMID 35450898
- [Background] Knight SR, Gupta RK, Ho A, Pius R, Buchan I, Carson G, Drake TM, Dunning J, Fairfield CJ, Gamble C, Green CA, Halpin S, Hardwick HE, Holden KA, Horby PW, Jackson C, Mclean KA, Merson L, Nguyen-Van-Tam JS, Norman L, Olliaro PL, Pritchard MG, Russell CD, Shaw CA, Sheikh A, Solomon T, Sudlow C, Swann OV, Turtle LCW, Openshaw PJM, Baillie JK, Docherty A, Semple MG, Noursadeghi M, Harrison EM; ISARIC Coronavirus Clinical Characterisation Consortium (ISARIC4C) Investigators; ISARIC4C investigators. Prospective validation of the 4C prognostic models for adults hospitalised with COVID-19 using the ISARIC WHO Clinical Characterisation Protocol. Thorax. 2022 Jun;77(6):606-615. doi: 10.1136/thoraxjnl-2021-217629. Epub 2021 Nov 22. PMID 34810237